CLINICAL TRIAL: NCT06842771
Title: Pain with Differing Intraperitoneal Washes At the End of Laparoscopic Gynecologic Surgery
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Tennessee (Other)
Responsible Party: Principal Investigator, John Schorge,MD, OB/GYN Chair and Professor, University of Tennessee
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 24-10173-FB
Record Dates: First submitted 2025-02-18; First posted 2025-02-24 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Laparoscopic Adnexal Surgery
Keywords: laparoscopic gynecologic surgery; adnexal laparoscopic surgery; ovarian laparoscopic surgery; fallopian tube laparoscopic surgery
MeSH Terms: interventions — Saline Solution

STUDY DESIGN:
Intervention Model Description: Prospective, single-blind, randomized clinical trial in participants who are undergoing planned, laparoscopic gynecologic surgery (adnexa only- the ovaries, fallopian tubes, and associated ligaments, vessels & connective tissue).
  A total of 96 women will be randomized to either the standard group or the comparator group. The control group (standard care) will receive an intraperitoneal wash with a fixed amount of saline. The experimental group (comparison treatment) will receive an intraperitoneal wash with an equal amount of pain medication.
  We have created a list of the participant counts;
  1. 8 blocks of 12, divided into 6 each: control and experimental.
  2. We have assigned a random number to each participant counted.
  3. Then, we have sorted each block by the random numbers. This gives a random ordering to the 6 control and 6 experimental participants within each block of 12. We will assign each participant to a condition in order of this sorted list.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Normal saline intraperitoneal wash post procedure (Active Comparator): The control group (standard care) will receive an intraperitoneal wash with a fixed amount of saline.
  Interventions: Other: Normal Saline (0.9% NaCl)
- Marcaine hydrochloride without epinephrine 0.5% intraperitoneal wash (Active Comparator): The experimental group (comparison treatment) will receive an intraperitoneal wash with 20 mL of Marcaine hydrochloride (bupivacaine) without epinephrine 0.5% at the end of surgery.
  Interventions: Drug: Marcaine hydrochloride without epinephrine 0.5%

INTERVENTIONS:
Other: Normal Saline (0.9% NaCl) — Women will undergo planned, laparoscopic gynecologic surgery with an intraperitoneal wash of 20 mL of saline (standard) at the end of the operation, prior to insufflation, release, and skin closure.
  The wash will be instilled into the peritoneal cavity and the surgical area (over the vaginal cuff and along the bilateral pelvic sidewalls to the paracolic gutters).
  All participants will rate their pain using a Visual Analogue Scale (VAS). The VAS is a numerical rating system where the scores range from zero (0) to ten (10), with zero indicating 'no pain at all' and ten indicating 'the worst possible pain'.
  Participants will be asked to rate their current level of pain and also report their current dosage of pain medication at the following intervals: pre-operatively, 2 hours post-operatively, and 24 hours post-operatively.
  Arms: Normal saline intraperitoneal wash post procedure
Drug: Marcaine hydrochloride without epinephrine 0.5% — Women will undergo planned, laparoscopic gynecologic surgery with an intraperitoneal wash of 20 mL Marcaine hydrochloride (bupivacaine) without epinephrine 0.5% (the comparator) at the end of the operation, prior to insufflation, release, and skin closure. The wash will be instilled into the peritoneal cavity and the surgical area (over the vaginal cuff and along the bilateral pelvic sidewalls to the paracolic gutters). All participants will rate their pain using a Visual Analogue Scale (VAS). The VAS is a numerical rating system where the scores range from zero (0) to ten (10), with zero indicating 'no pain at all' and ten indicating 'the worst possible pain'. Participants will be asked to rate their current level of pain and also report their current dosage of pain medication at the following intervals: pre-operatively, 2 hours post-operatively, and 24 hours post-operatively.
  Arms: Marcaine hydrochloride without epinephrine 0.5% intraperitoneal wash

SUMMARY:
We hypothesize that instilling intraperitoneal Marcaine (without epinephrine) at the end of a non-total laparoscopic gynecologic surgery (adnexa only, which includes the ovaries, fallopian tubes, and associated ligaments, vessels, and connective tissue) will result in less pain and reduced opioid use postoperatively.

DETAILED DESCRIPTION:
Minimally invasive gynecologic surgery has been shown to reduce postoperative pain, length of hospital stay, and prescription opioid use when compared to open procedures. However, postoperative abdominal pain is still significant, and the ways in which this pain can be reduced requires further exploration.

It is standard procedure to inject the surgical incision sites with long-acting analgesics such as Marcaine or Ropivacaine. However, intraperitoneal instillation of these pain medications and their effect on postoperative pain and prescription opioid use has only minimally been explored thus far.

In a retrospective cohort study, the effectiveness of administering intraperitoneal bupivacaine on decreasing postoperative pain in patients undergoing minimally invasive gynecologic surgery was evaluated. For the 130 patients included in the study, those who received the intraperitoneal bupivacaine "had lower median narcotic use on the day of surgery and the first postoperative day, compared with those who did not receive intraperitoneal bupivacaine".

Given these results, we believe that it will be beneficial to include the use of intraperitoneal anesthetics for patients receiving laparoscopic gynecologic surgery (adnexa only, which includes the ovaries, fallopian tubes, and associated ligaments, vessels, and connective tissue).

Marcaine hydrochloride (bupivacaine) without epinephrine 0.5% was chosen for this study because this was used in previous studies, and it is used for analgesia at the trocar incisions during the laparoscopic procedure. The extra Marcaine hydrochloride (bupivacaine) without epinephrine 0.5% will, therefore, be available for use instead of being discarded. The use of Marcaine hydrochloride (bupivacaine) without epinephrine 0.5% will not incur any additional cost. Similarly, normal saline is used routinely during these types of surgical procedures, is available post-operatively for use as an intraperitoneal wash instead of being discarded. The participants will be randomized to Marcaine hydrochloride (bupivacaine) without epinephrine 0.5% or normal saline.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older
* Undergoing planned laparoscopic adnexal surgery as a day surgery procedure; The surgical site is the "adnexa" which contains the ovaries, fallopian tubes, and associated ligaments, vessels, and connective tissue. The "adnexa" does not include the uterus.
* BMI 55.0 or less

Exclusion Criteria:

* Under age 18
* Undergoing a non-laparoscopic unplanned surgical procedure Patients having a laparoscopic partial or complete removal of the uterus, a hysterectomy, will NOT be included in this study population for enrollment.
* septicemia
* severe hemorrhage
* severe hypotension or shock
* arrhythmias
* known hypersensitivity to bupivacaine or to any other local anesthetic agent
* local infection at the injection site

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
subjective pain scores | At approximately 24 hours after surgery completion
  At approximately 24 hours after surgery completion, we will contact the participant in person if still hospitalized, or via telephone if discharged home, to ask what their pain level is (utilizing the VAS) and how many opioid tablets (mg dosage and number) they have used since hospital discharge.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Tennessee Health Science Center, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No